CLINICAL TRIAL: NCT00607230
Title: Determination of Dosing and Frequency of BCG Administration Necessary to Alter T-Lymphocyte Profiles in Type I Diabetics
Brief Title: Determination of Dosing and Frequency of BCG Administration to Alter T-Lymphocyte Profiles in Type I Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David M. Nathan, MD, Director, Diabetes Center, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007p-001347
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; immune modulation; cure; autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E (Experimental): BCG vaccination
  Interventions: Biological: BCG
- P (Placebo Comparator): Saline vaccination
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: BCG — BCG vaccination at 0 and 4 weeks
  Arms: E
Biological: Saline — Saline vaccination at 0 and 4 weeks
  Arms: P

SUMMARY:
Type 1 diabetes is caused by an autoimmune destruction of the insulin producing cells of the pancreas. The investigators have discovered the specific autoimmune cells responsible for destroying the insulin-producing cells in an animal model of type 1 diabetes, and the means of destroying those cells.

DETAILED DESCRIPTION:
The investigators are now aiming to use a similar strategy (vaccination with BCG, the vaccine used world-wide to protect against tuberculosis) in human type 1 diabetes to see if the abnormal immune cells can be depleted. This is the first step in trying to cure established type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria (Type 1 diabetic subjects):

* Type 1 diabetes treated continuously with insulin from time of diagnosis
* Age 18-55
* Anti-GAD positive
* HIV antibody negative
* Normal CBC
* Negative intermediate PPD test performed and read by study staff
* HCG Negative (females)

Exclusion Criteria Type 1 diabetic subjects):

* History of chronic infectious disease, such as HIV
* History of tuberculosis, TB risk factors, or history of + PPD, or BCG vaccination
* Treatment with glucocorticoids (other than intermittent nasal steroids) or disease or condition likely to require steroid therapy
* Other conditions or treatments associated with increased risk of infections such as patients with previous history of severe burns, or treatment with immunosuppressive medications of any type (e.g. imuran, methotrexate, cyclosporine, etanercept, infliximab) for any reason
* Current treatment with aspirin > 160 mg/day or chronic, daily NSAIDs
* Fasting or stimulated (1 mg glucagon stimulation test) c-peptide > 0.2 pmol/mL
* History of keloid formation
* HbA1c > 8.0%
* History or evidence of chronic kidney disease (serum creatinine > 1.5 mg/dL)
* History of proliferative diabetic retinopathy that has not been treated with laser therapy
* Pregnant or not using acceptable birth control
* Living with someone who is immunosuppressed and/or at high risk for infectious diseases (for example HIV+ or taking immunosuppressive medications for any reason).

Inclusion Criteria (Control Non-diabetic Subjects):

* Age 18-45

Exclusion Criteria (Control Non-diabetic Subjects):

* History of autoimmune diseases or diabetes
* History of HIV History of autoimmune disease or type 1 diabetes (use of insulin continuously since diagnosis) in first degree family members

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
concentration of autoreactive t-cells | Measured weekly in first 8 weeks, then every other week for weeks 8-12

SECONDARY OUTCOMES:
Concentration of TNF, TNF-receptors, other cytokines, and c-peptide levels | Weekly for first 8 weeks, then every other week for weeks 8-12

CONTACTS AND LOCATIONS:
Overall Officials: David M Nathan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Diabetes Research Center at Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Faustman DL, Wang L, Okubo Y, Burger D, Ban L, Man G, Zheng H, Schoenfeld D, Pompei R, Avruch J, Nathan DM. Proof-of-concept, randomized, controlled clinical trial of Bacillus-Calmette-Guerin for treatment of long-term type 1 diabetes. PLoS One. 2012;7(8):e41756. doi: 10.1371/journal.pone.0041756. Epub 2012 Aug 8. PMID 22905105